CLINICAL TRIAL: NCT04555811
Title: FATE FT596 With Rituximab as Relapse Prevention in High Risk Patients After Autologous Hematopoietic Stem Cell Transplantation for Non-Hodgkin Lymphoma
Brief Title: FT596 With Rituximab as Relapse Prevention After Autologous HSCT for NHL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2019LS230; P01CA111412 (NIH)
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Results first posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: NHL; Non Hodgkin Lymphoma; Diffuse Large B Cell Lymphoma; High-grade B-cell Lymphoma
Keywords: auto HSCT; Stem cell transplantation; Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma | interventions — Rituximab

STUDY DESIGN:
Intervention Model Description: Patients are enrolled in cohorts of 3 starting at Dose Level 1. There are three dose escalating doses of FT596. A minimum of 28 days will separate each cohort. For Dose Level 1 a minimum of 28 days will separate each patient to assess for dose limiting toxicity (DLT). In subsequent cohorts, the 1st and 2nd patient will be separated by at least 28 days and at least 14 days will separate the 2nd and 3rd patient.
  Each new cohort of three patients will be sequentially assigned to the most appropriate dose based on the updated toxicity probabilities under the continuous reassessment method (CRM), and the MTD will be identified when the total sample size of 18 is exhausted or 6 patients are sequentially enrolled at the same dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- FT596 + Rituximab Dose Level 1: 9x10^7 cells/dose (Experimental): Up to three sequential FT596 dose levels are planned for Day 30 administration: (Dose Level 1: 9x10^7 cells/dose, Dose Level 2: 3x10^8 cells/dose, Dose Level 3: 9x10^8 cells/dose with a Dose Level -1: 3x10^7 cells/dose tested only if dose limiting toxicity events (DLT) occur at dose level 1).The maximum tolerated dose will be determined by using a modified continual reassessment method (CRM).
  Interventions: Drug: FT596; Drug: Rituximab
- FT596 + Rituximab Dose Level 2: 3x10^8 cells/dose (Experimental): Up to three sequential FT596 dose levels are planned for Day 30 administration: (Dose Level 1: 9x10^7 cells/dose, Dose Level 2: 3x10^8 cells/dose, Dose Level 3: 9x10^8 cells/dose with a Dose Level -1: 3x10^7 cells/dose tested only if dose limiting toxicity events (DLT) occur at dose level 1).The maximum tolerated dose will be determined by using a modified continual reassessment method (CRM).
  Interventions: Drug: FT596; Drug: Rituximab
- FT596 + Rituximab Dose Level 3: 9x10^8 cells/dose (Experimental): Up to three sequential FT596 dose levels are planned for Day 30 administration: (Dose Level 1: 9x10^7 cells/dose, Dose Level 2: 3x10^8 cells/dose, Dose Level 3: 9x10^8 cells/dose with a Dose Level -1: 3x10^7 cells/dose tested only if dose limiting toxicity events (DLT) occur at dose level 1).The maximum tolerated dose will be determined by using a modified continual reassessment method (CRM).
  Interventions: Drug: FT596; Drug: Rituximab

INTERVENTIONS:
Drug: FT596 — FT596 is given 2-3 days after rituximab; however, it may be delayed for up to 7 days until all rituximab infusion related toxicities resolve to ≤Grade 1.
Drug: Rituximab — Rituximab 375 mg/m^2 is administered as an IV infusion per institutional standard of care and package insert on 2-3 days (48 to 72 hours) prior to the FT596 infusion
  Other Names: Rituxan

SUMMARY:
This is a Phase I multi-center study to evaluate the safety of FT596 when given with rituximab as relapse prevention in patients who have undergone an autologous hematopoietic stem cell transplant (auto-HSCT) for diffuse large or high-grade B cell lymphoma.

DETAILED DESCRIPTION:
This study uses a single dose of the investigational product FT596 in the early post-transplant period. Rituximab or an FDA approved by biosimilar including Rituxan®, Truxima®, and Ruxience™ is given 48 to 72 hours prior to FT596. The goal of this study is to 1) establish a maximum tolerated dose (MTD) of FT596 when given 30 days after transplant and 2) to confirm the MTD and safety of giving a single dose of FT596 at Day 7 post-transplant starting at one dose level below the MTD identified at Day 30.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diffuse large B cell lymphoma or aggressive (high-grade) B-cell lymphoma for which an autologous stem cell transplant is planned or recently completed
* High risk for relapse defined as at least one of the below:

  * Primary induction failure (no complete or partial remission at any point after diagnosis
  * Initial remission duration < 12 months
  * Lack of complete metabolic (PET scan) response after 2-3 cycles of salvage chemotherapy
  * Evidence of c-myc and bcl-2 and/or bcl-6 re-arrangement (double hit or triple hit lymphoma)
  * Age-adjusted IPI 2-3 at relapse
* Age 18 years or older at the time of signing consent.
* Agrees to use adequate contraception (or evidence of sterility) for at least 12 months after the last dose of rituximab.
* Agrees and signs the separate consent for up to 15 years of follow-up (Long-term Follow-up study CPRC#2020LS052)
* Provides voluntary written consent prior to the performance of any research related activities.

Exclusion Criteria:

* Receipt of any investigational therapy within 28 days prior to the first dose of FT596 or planned use of an investigational therapy during the first 100 days after transplant
* Planned post-transplant irradiation prior to Day +100
* Seropositive for HIV, active Hepatitis B or C infection with detectable viral load by PCR
* Body weight <50kg
* Known allergy to the following FT596 components: albumin (human) or DMSO
* Unable to receive rituximab

Post-HSCT Reconfirmation of eligibility

* No life-threatening medical issues (i.e. ongoing Grade 4 adverse events) where, in the opinion of the treating investigator, use of FT596 is not in the patient's best interest.
* No active uncontrolled infection.
* Adequate organ function post-transplant including:

  * alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤5 x ULN (Grade 2 CTCAE v5)
  * total bilirubin ≤1.5 x ULN (Grade 1 CTCAE v5)
  * serum creatinine ≤1.5 x ULN (Grade 1 CTCAE v5)
  * oxygen saturation ≥93% on room air
* For Day 30 dosing only - CBC requirement consistent with engraftment (ANC>500, platelet>20,000 without transfusion support within previous 7 days). There are no CBC parameters for Day 7 dosing.
* No requirement for systemic immunosuppressive therapy (> 5mg prednisone daily) during the FT596 dosing period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Veronika Bachanova, MD, PhD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FT596 + Rituximab Dose Level 1: 9x10^7 Cells/Dose | FT596 + Rituximab Dose Level 2: 3x10^8 Cells/Dose | FT596 + Rituximab Dose Level 3: 9x10^8 Cells/Dose
Started | 3 | 3 | 1
Completed | 3 | 3 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FT596 + Rituximab Dose Level 1: 9x10^7 Cells/Dose | FT596 + Rituximab Dose Level 2: 3x10^8 Cells/Dose | FT596 + Rituximab Dose Level 3: 9x10^8 Cells/Dose | Total
Number analyzed (Participants) | 3 | 3 | 1 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 1 | 5
  >=65 years | 1 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1
  Male | 2 | 3 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 1 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 2 | 1 | 5
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Dose Limiting Toxicity Events
Description: The component I design (FT596 on day 30) will continue until the MTD is declared or until the first dose is declared to be above MTD. The component I dose limiting toxicity (DLT) is defined as any of the following events within 28 days after the FT596 dosing based on CTCAE v5:Grade 4 hematologic toxicity lasting > 7 days ,Grade 4 non-hematologic toxicity ,Grade ≥3 Infusion Related Reaction, Grade 2 acute GVHD that requires steroid therapy >7 days or progression after 3 days of steroids or has partial response after 14 days of treatment, Grade ≥3 acute GVHD, Grade 4 cytokine release syndrome (CRS), Grade 3 CRS that does not resolve to < Grade 2 in 72 hours, Grade 3 neurotoxicity, Grade 3 organ toxicity involving vital organs, Any Grade 3 non-hematological toxicity that does not resolve to ≤Grade 2 within 72 hours
Time Frame: 28 Days Post FT596 infusion
Measure: Count of Participants; unit: Participants
Arm/Group | FT596 + Rituximab Dose Level 1: 9x10^7 Cells/Dose | FT596 + Rituximab Dose Level 2: 3x10^8 Cells/Dose | FT596 + Rituximab Dose Level 3: 9x10^8 Cells/Dose
Number analyzed (Participants) | 3 | 3 | 1
Participants | 0 | 0 | 0

2. Secondary Outcome: Number of Participants Experiencing Adverse Events
Description: Number of participants experiencing adverse events related to FT596 post auto-HSCT in combination with rituximab
Time Frame: 1 year post FT596 infusion
Measure: Number; unit: participants
Arm/Group | FT596 + Rituximab Dose Level 1: 9x10^7 Cells/Dose | FT596 + Rituximab Dose Level 2: 3x10^8 Cells/Dose | FT596 + Rituximab Dose Level 3: 9x10^8 Cells/Dose
Number analyzed (Participants) | 3 | 3 | 1
participants | 3 | 0 | 1

3. Secondary Outcome: Percentage of Participants With Relapse/Progression
Description: Percentage of participants experiencing progression or relapse at 12 months post auto HSCT
Time Frame: 1 year post auto HSCT
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FT596 + Rituximab Dose Level 1: 9x10^7 Cells/Dose | FT596 + Rituximab Dose Level 2: 3x10^8 Cells/Dose | FT596 + Rituximab Dose Level 3: 9x10^8 Cells/Dose
Number analyzed (Participants) | 3 | 3 | 1
Percentage of participants | 67 [22 to 100] | 33 [0 to 77] | 0 [0 to 100]

4. Secondary Outcome: Number of Participants Experiencing Non-relapse Mortality Incidents at 100 Days Post HSCT
Description: Number of participants experiencing non-relapse mortality at 100 days post auto-HSCT.
Time Frame: 100 days post HSCT
Measure: Count of Participants; unit: Participants
Arm/Group | FT596 + Rituximab Dose Level 1: 9x10^7 Cells/Dose | FT596 + Rituximab Dose Level 2: 3x10^8 Cells/Dose | FT596 + Rituximab Dose Level 3: 9x10^8 Cells/Dose
Number analyzed (Participants) | 3 | 3 | 1
Participants | 0 | 0 | 0

5. Secondary Outcome: Percentage of Non-relapse Mortality Incidents at One Year Post HSCT
Description: Percentage of participants experiencing non-relapse mortality at one year post auto-HSCT.
Time Frame: one year post auto-HSCT
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FT596 + Rituximab Dose Level 1: 9x10^7 Cells/Dose | FT596 + Rituximab Dose Level 2: 3x10^8 Cells/Dose | FT596 + Rituximab Dose Level 3: 9x10^8 Cells/Dose
Number analyzed (Participants) | 3 | 3 | 1
Percentage of participants | 67 [5 to 95] | 100 [0 to 100] | 100 [0 to 100]

6. Secondary Outcome: Progression-Free Survival 12 Months Post Auto-HCT
Description: Progression-Free Survival 12 Months Post Auto-HCT
Time Frame: 12 Months Post Auto-HCT
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FT596 + Rituximab Dose Level 1: 9x10^7 Cells/Dose | FT596 + Rituximab Dose Level 2: 3x10^8 Cells/Dose | FT596 + Rituximab Dose Level 3: 9x10^8 Cells/Dose
Number analyzed (Participants) | 3 | 3 | 1
Percentage of participants | 33 [1 to 77] | 67 [5 to 95] | 100 [0 to 100]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | FT596 + Rituximab Dose Level 1: 9x10^7 Cells/Dose | FT596 + Rituximab Dose Level 2: 3x10^8 Cells/Dose | FT596 + Rituximab Dose Level 3: 9x10^8 Cells/Dose
All-Cause Mortality (participants affected / at risk) | 2/3 | 3/3 | 1/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 0/3 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FT596 + Rituximab Dose Level 1: 9x10^7 Cells/Dose (N=3) | FT596 + Rituximab Dose Level 2: 3x10^8 Cells/Dose (N=3) | FT596 + Rituximab Dose Level 3: 9x10^8 Cells/Dose (N=1)
Lymphocyte count decreased (Investigations) | 1 (9) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (4) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (5) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (3) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/11/NCT04555811/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT04555811/ICF_001.pdf